CLINICAL TRIAL: NCT02695225
Title: Tobacco Cessation Interventions With Ohio Appalachian Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary Ellen Wewers, Professor Emerita, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008H0298; R01CA129771 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lay-led tobacco abstinence (Other): Each intervention visit, which lasts an average of 30 minutes, will be delivered face-to-face in a mutually agreed upon convenient location (e.g. participant's home, county extension office). All behavioral and pharmacological intervention strategies will be delivered by the lay educator, with supervision by the county nurse (assigned by county with no overlap between conditions). As recommended by the USPHS guideline, all participants will set a 'quit date' and receive identical behavioral and pharmacological treatment throughout the intervention.
  Interventions: Behavioral: Lay-led tobacco abstinence
- Lay-led promotion of Ohio Quit Line (Other): Each participant will be given print information about the Ohio Tobacco QUIT LINE (1-800-QUIT-NOW) and encouraged to call for proactive telephone counseling and free NRT. Proactive telephone counseling and NRT administration will be provided by a QUIT LINE counselor, using their standard protocol.
  Interventions: Behavioral: Lay-led promotion of Ohio Quit Line

INTERVENTIONS:
Behavioral: Lay-led tobacco abstinence — Lay-led tobacco abstinence: Each intervention visit, which lasts an average of 30 minutes, will be delivered face-to-face in a mutually agreed upon convenient location (e.g. participant's home, county extension office). All behavioral and pharmacological intervention strategies will be delivered by the lay educator, with supervision by the county nurse (assigned by county with no overlap between conditions). As recommended by the USPHS guideline, all participants will set a 'quit date' and receive identical behavioral and pharmacological treatment throughout the intervention.
  Arms: Lay-led tobacco abstinence
Behavioral: Lay-led promotion of Ohio Quit Line — Lay-led promotion of Ohio Quit Line (control condition): Each participant will be given print information about the Ohio Tobacco QUIT LINE (1-800-QUIT-NOW) and encouraged to call for proactive telephone counseling and free NRT. Proactive telephone counseling and NRT administration will be provided by a QUIT LINE counselor, using their standard protocol.
  Arms: Lay-led promotion of Ohio Quit Line

SUMMARY:
Tobacco use remains a significant public health problem and is increasingly prevalent among vulnerable groups. Appalachians have a high prevalence of tobacco use and are at increased risk for tobacco-attributable diseases. The efficacy of a scientifically valid tobacco cessation treatment delivered to Appalachian smokers remains untested. Also, little is known about the association of social-contextual factors that may modify or mediate the success of an intervention. These factors may be of particular relevance among disadvantaged smokers. Geographical patterns of tobacco exposure may also influence one's ability to quit, especially in pro- tobacco regions like Appalachia. The purposes of this application are to: 1) evaluate the efficacy of a lay-led (LL) intervention in promoting long term abstinence from tobacco; and 2) examine the association between 12 month abstinence and selected individual, interpersonal, organizational, neighborhood and community, and societal factors among adult Appalachian tobacco users exposed to a tobacco cessation intervention. A third aim is exploratory and includes the characterization of activity patterns using space-time measures among adult Appalachian tobacco users exposed to a tobacco cessation intervention. Using a group randomized trial design, 707 Appalachian residents from 6 intervention and 6 control counties will be randomly assigned by county to receive the LL intervention or a control condition which includes proactive telephone counseling via the Ohio Quit Line. LL group participants will receive face-to-face counseling, supervised by a county health department nurse, and delivered by a trained lay educator. A county Extension agent will assist with recruitment and retention efforts in this project. Social-contextual factors will be assessed at a baseline interview administered to all participants. Space-time activity geographical patterns of pro- and anti-tobacco exposures, or features, will be described among selected participants in four counties during weeks 1, 6 and 12 of treatment. At end of treatment and 6 and 12 months, LL and control group participants will be reassessed for tobacco use via self-report and cotinine-validation. Secondary analyses will explore differential trends over time between the two arms of the study. In a subset of the sample, pro- and anti-tobacco exposures will be estimated during weeks 1, 6 and 12 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years and older
* Current self-reported use of tobacco on a daily basis
* Resident of one of the 12 participating counties
* Absence of clinical condition that contraindicates use of over-the-counter NRT, including: severe arrhythmias, severe angina, or myocardial infarction within the previous 4 weeks
* If female, non-pregnant, as confirmed by urine human chorionic gonadotropin (HCG) test

Only one member per household will be enrolled. If more than one member is interested, the member whose birthday is closest to date of enrollment will be chosen. Once 12 month data collection is completed for the participant, cessation materials/referral to the Ohio Quit Line will be offered to other interested family member(s).

Exclusion Criteria:

* Under 18 years of age
* Non-daily use of tobacco (self-reported)
* Not a resident of one of the 12 participating counties
* Presences of clinical condition that contraindicates use of over-the-counter NRT, including: severe arrhythmias, severe angina, or myocardial infarction within the previous 4 weeks
* If female, pregnant, as confirmed by urine human chorionic gonadotropin (HCG) test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2010-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Self-reported tobacco abstinence in past 7 days as confirmed by saliva cotinine concentration < 15ng/ml | 12 months
  At the 12 month time point, tobacco abstinence (past 7 days) will be assessed using self-reported data. Saliva cotinine concentration of less than 15ng/ml will confirm as abstinence.